CLINICAL TRIAL: NCT04943341
Title: Eco-guided Treatment With Triamcinolone-Acetonide in the Treatment of Medial Plica Syndrome - A Pilot Study
Brief Title: Evaluation of the Triamcinolone -Acetonide Therapy for the Treatment of the Medial Plica Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PLICA
Record Dates: First submitted 2021-05-17; First posted 2021-06-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Medial Plica Syndrome
Keywords: medial plica syndrome; medial plica; knee; Pilot study; Triamcinolone Acetonide; injection treatment

STUDY DESIGN:
Intervention Model Description: The pilot study will be include a single group of 30 patience affected by the medial plica syndrome. Patients will be treated with an eco-guided injection of Triamcinolone-Acetonide and will be evaluated clinical and radiological outcomes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Eco-guided Triamcinolone-Acetonide injection (Experimental): Patients affected by medial plica syndrome will be treated with an eco-guided injection of Triamcinolone-Acetonide.
  Interventions: Procedure: Eco-guided Triamcinolone-Acetonide injection

INTERVENTIONS:
Procedure: Eco-guided Triamcinolone-Acetonide injection — The treatment consists in injecting 1 ml of Kenacort (corresponding to 40 mg of Triamcinolone Acetonide) diluted in about 1 ml of local anesthetic (Lidocaine) directly into the medial fold of the knee. Through an ultrasound guidance with "in plane" technique, the flute beak of the needle will be positioned between the two sheets of the synovial fold and the injection will be performed.

SUMMARY:
The aim of this pilot study is to evaluate the clinical and radiological outcomes (ultrasound and MRI) for a treatment utilized in the medial plica syndrome resistant to conservative therapy. Will be evaluated an intra-plica ultrasound-guided injections of Triamcinolone-Acetonide and lidocaine percutaneously, and associated rehabilitation therapy. The aim of the study will be to evaluate the efficacy and safety of the injection procedure by revealing clinical improvement and monitoring the incidence of adverse events following treatment.

DETAILED DESCRIPTION:
30 patients affected by the medial plica syndrome will be included in a pilot study in which one will be evaluated the effect of treatment with Triamcinolone-Acetonide and Lidocaine, injected intraplical with an ultrasound-guided procedure. For evaluating the treatment, will be considered functional and pain outcomes. Patients will be evaluated before treatment by a clinical, an MRI and an ultrasound examination. After the injection, they will be followed up at 1, 3, 6 and 12 months. At the 1 and 3 month FU visits patients will be evaluated by an ultrasound examination and at the 6 month FU they will be evaluated by an MRI examination.

ELIGIBILITY:
Inclusion Criteria:

1. Ultrasonographic and/or MRI signs of medial plica pathology;
2. VAS pain 4-8 at time of inclusion;
3. Failure, defined as the persistence of symptomatology, after at least one course of conservative treatment of at least 6 weeks (rest and drug treatment, physiotherapy);
4. Ability and consent of patients to actively participate in clinical follow-up;

Exclusion Criteria:

1. BMI > 35;
2. Patients with: rheumatic diseases, diabetes, infectious processes, epilepsy, severe stage osteoporosis
3. Patients undergoing intra-tendon infiltration of other substance within the previous 6 months;
4. Patients undergoing surgery on the affected knee within the previous 12 months;
5. Patients undergoing femoro- patellar joint stabilization surgery to the affected knee;
6. Trauma to the affected knee within the past 6 months;
7. Episodes of patellar dislocation and subluxation to the affected knee;
8. State of immunodepression;
9. Ongoing systemic inflammatory diseases (stabilized outcomes of these diseases are not considered absolute contraindications).
10. Contraindications to use or hypersensitivity to the active ingredient (Triamcinolone Acetonide) or to the excipients (sodium chloride, benzyl alcohol, sodium carboxymethylcellulose, polysorbate 80 and water for injectable preparations)found within Kenacort as per the product package insert;

12. Contraindications or hypersensitivity to the active ingredient of the local anesthetic (Lidocaine) or their excipients; 13. Pregnancy or lactation status or intention to become pregnant during the period of study participation. In particular, in the case of a suspected pregnancy , this will be excluded by serological testing (hCG).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2024-09-16 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
KUJALA Scale (Kujala Anterior Knee Pain Scale (AKPS | 6 months FU
  This is a patient-reported assessment of patellofemoral disorders that evaluates subjective symptoms and functional limitations. The evaluation consist of 13 questions with a total score of 100 points.

SECONDARY OUTCOMES:
KOOS (Knee Injury and Osteoarthritis Outcome Score) | baseline, 1 month, 3 months, 6 and 12 months FU
  KOOS SCORE consists of 5 subscales and covers: pain (9 items), symptoms (7 items, two of which are related to stiffness), functions and activities of daily living (17 items), physical function, sports and leisure activities (5 items) and quality of life in relation to the knee (4 items).
VAS (Visual Analogue Scale) | baseline, 1 month, 3 months, 6 and 12 months FU
  VAS is a visual analogue scale consisting of a range scale (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable
Patient Acceptable Symptom State (PASS) | baseline, 1 month, 3 months, 6 and 12 months, 24 months FU
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no".
Ultrasound assessment | baseline, 1 month, 3 months FU
  This examination is useful to evaluate the evolution of plica thickness;
MRI assessment | baseline, 6 months FU
  This assessment is useful for evaluating plica retraction
Final treatment opinion | 24 months follow-up
  The patient should indicate satisfaction and relative degree with treatment at the end of the clinical trial (24 months follow-up). All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "much better", "somewhat better", "no change", "a little worse", "much worse".
Patient Rehabilitation Monitoring | 12 months follow-up
  The patient will be asked if he/she performs the planned rehabilitation activity for the 12 weeks following treatment. All patients will be able to answer "yes"or "no" regarding the rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Andriolo, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bellary SS, Lynch G, Housman B, Esmaeili E, Gielecki J, Tubbs RS, Loukas M. Medial plica syndrome: a review of the literature. Clin Anat. 2012 May;25(4):423-8. doi: 10.1002/ca.21278. PMID 22331585
- [Background] Dupont JY. Synovial plicae of the knee. Controversies and review. Clin Sports Med. 1997 Jan;16(1):87-122. doi: 10.1016/s0278-5919(05)70009-0. PMID 9012563
- [Background] Jee WH, Choe BY, Kim JM, Song HH, Choi KH. The plica syndrome: diagnostic value of MRI with arthroscopic correlation. J Comput Assist Tomogr. 1998 Sep-Oct;22(5):814-8. doi: 10.1097/00004728-199809000-00028. PMID 9754123
- [Background] Amatuzzi MM, Fazzi A, Varella MH. Pathologic synovial plica of the knee. Results of conservative treatment. Am J Sports Med. 1990 Sep-Oct;18(5):466-9. doi: 10.1177/036354659001800503. PMID 2252085
- [Background] Rovere GD, Adair DM. Medial synovial shelf plica syndrome. Treatment by intraplical steroid injection. Am J Sports Med. 1985 Nov-Dec;13(6):382-6. doi: 10.1177/036354658501300603. PMID 4073344
- [Background] Collins NJ, Prinsen CA, Christensen R, Bartels EM, Terwee CB, Roos EM. Knee Injury and Osteoarthritis Outcome Score (KOOS): systematic review and meta-analysis of measurement properties. Osteoarthritis Cartilage. 2016 Aug;24(8):1317-29. doi: 10.1016/j.joca.2016.03.010. Epub 2016 Mar 21. PMID 27012756
- [Background] Delgado DA, Lambert BS, Boutris N, McCulloch PC, Robbins AB, Moreno MR, Harris JD. Validation of Digital Visual Analog Scale Pain Scoring With a Traditional Paper-based Visual Analog Scale in Adults. J Am Acad Orthop Surg Glob Res Rev. 2018 Mar 23;2(3):e088. doi: 10.5435/JAAOSGlobal-D-17-00088. eCollection 2018 Mar. PMID 30211382